CLINICAL TRIAL: NCT05054270
Title: Efficacy of Lung Ultrasound in Monitoring Fluid Resuscitation in Trauma Patients
Brief Title: Efficacy of Lung Ultrasound in Monitoring Fluid Resuscitation in Chest Trauma Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Yassien Mahmoud Ahmed, Emergency medicine resident physician, Assiut University
Other Study IDs: Chest US in lung contusion
Record Dates: First submitted 2021-06-02; First posted 2021-09-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2021-07

CONDITIONS: Contusions Pulmonary; Lung Injury; Chest Trauma; Fluid Overload Pulmonary Edema
MeSH Terms: conditions — Lung Injury; Thoracic Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chest examination with Ultrasound device — Chest examination with Ultrasound device

SUMMARY:
Efficacy of Lung ultrasound in monitoring fluid resuscitation in chest trauma patients with lung contusions

DETAILED DESCRIPTION:
Trauma is a public health problem, associated to high morbidity and mortality, In Egypt the mortality from road traffic crashes is about 12000 victims per year.

* Chest trauma represents from 10% to 15% of the total number of traumas worldwide.

According to ATLS protocol , early diagnosis and management of Chest trauma are essential. *Pulmonary contusion is found in 30-75% of cases of chest injury.

* point of care Ultrasound (POCUS) is Now a corner stone in Emergency management it can predict lung contusions within the first 72 hours after trauma.
* Recently, LUS Play a major role in assessment of the volume status in Trauma patients.
* B-lines score (BLS) has been validated as a lung ultrasound quantification of pulmonary congestion.The sum of all B-lines yields a score, B-lines score (BLS), which assess the degree of lung contusion. So that LUS may provide a valuable safety threshold to conduct fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* chest trauma patients either with or without other injuries.
* Any patient with either blunt or penetrating chest trauma.

Exclusion Criteria:

* - Patients in cardiac arrest.
* Patient refusal to participate
* Pregnant females.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is an observational study that will be conducted on patients admitted with chest trauma in Assuit or Alexandria Main University Hospitals after obtaining their or their next of kin consent to participate in the study without affecting their course of treatment according to permission obtained from ethical committee of faculty of medicine in Assiut and Alexandria universities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with lung contusion | Upto 24 hours after trauma
  Pulmonary edema will be detected by B_lines trauma patients with lung contusions

SECONDARY OUTCOMES:
Clinical correlation between Type & volume of Fluid & occurance of pulmonary edema. Correlation between severity of pulmonary lung contusion & The final disposition of the patients whatever (OR _another department _death….. etc) upto 24hr. | For first 24 hours after trauma
  Follow up on degree of contusions after fluid resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ullman EA, Donley LP, Brady WJ. Pulmonary trauma emergency department evaluation and management. Emerg Med Clin North Am. 2003 May;21(2):291-313. doi: 10.1016/s0733-8627(03)00016-6. PMID 12793615
- [Background] Miller DL, Mansour KA. Blunt traumatic lung injuries. Thorac Surg Clin. 2007 Feb;17(1):57-61, vi. doi: 10.1016/j.thorsurg.2007.03.017. PMID 17650697
- [Background] Cohn SM. Pulmonary contusion: review of the clinical entity. J Trauma. 1997 May;42(5):973-9. doi: 10.1097/00005373-199705000-00033. PMID 9191684